CLINICAL TRIAL: NCT05721820
Title: Aortic Cross-clamp and Opening After Transcatheter Aortic Valve Implantation: a Real Issue?
Status: Completed | Type: Observational
Sponsor: Michele De Bonis (Other)
Responsible Party: Sponsor-Investigator, Michele De Bonis, Chief of Cardiac Surgery of Advanced and Research Therapies, Ospedale San Raffaele
Organization: Ospedale San Raffaele (Other)
Other Study IDs: AXC-TAVI
Record Dates: First submitted 2023-01-26; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Aortic Stenosis
Keywords: TAVR
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: TAVR — Transcatheter aortic valve replacement

SUMMARY:
Since its first clinical introduction by Alan Cribier in 2002, transcatheter aortic valve implantation has become the treatment of choice for severe aortic stenosis in high-risk and elderly patients. In such a population, cardiac surgery after TAVI is seldom performed (<1%), and only in cases of life-threatening complications such as device embolization, heart rupture, aortic dissection, endocarditis, etc.

* State-of-the-art Nowadays, patients submitted to TAVI are getting younger, with lower surgical risk and longer life-expectancy, and their number is continuously increasing . As a consequence, the number of patients treated with TAVI who will require subsequent cardiac surgery will also expand, both acutely (due to the above-mentioned complications) and during follow-up (due to late endocarditis, valve degeneration and other non-aortic indications).
* Previous informations Despite cardiac surgery after TAVI has been already performed several times across the world without documented issues in regard to aortic cross-clamp and aortotomy, it has been long debated whether the presence of TAVI devices with a tall stent frame in the ascending aorta may theoretically jeopardize the ability of surgeons to clamp and open the aorta. No specific data is yet available in regard to the existence and the incidence of such issue.
* Ethical issues Not present.

Aim of the study The aim of this study was to assess the anatomical feasibility of surgical aortic cross-clamp and aortotomy after TAVI based on post-TAVI computed tomographies (CT).

Study design This study enrolled patients who underwent TAVI in three high-volume centers (San Raffaele University Hospital in Milan - Italy, Rigshospitalet Univeristy Hospital in Copenhagen - Denmark, Semmelweiss University in Budapest - Hungary) between October 2008 and May 2017.

117 CT acquired after TAVI procedures that were cardiac-gated and included the aortic arch into the field of view were retrospectively reviewed. 11 patients of San Raffaele Hospital will be involved.

Reasons for post-TAVI acquisition were: participation into a clinical study with a previous Ethical Committee approval (91.4% n = 107); residual aortic regurgitation assessment for Valve-in-Valve evaluation (6.0% n = 7); TAVI complication assessment (ventricular septum defect 1.7% n = 2, left ventricular outflow tract obstruction 0.9% n = 1). Median time of CT acquisition after TAVI was 451 [290-780] days.

As per study design, only TAVI devices with a long stent were assessed: CoreValve (Medtronic Inc., MN, USA) n = 82 (size 26 n = 23; size 29 n = 48; size 31 n = 11); CoreValve Evolut R (Medtronic Inc., MN, USA) n = 19 (size 23 n = 1; size 26 n = 7; size 29 n = 10; size 34 n = 1); Portico (Abbott, IL; USA) n = 16 (size 25 n = 9; size 27 n = 4; size 29 n = 3). Acurate Neo device (Boston Scientific, MA, USA, former Symetis) presents three stabilization arches in the ascending aorta which differ this prosthesis from the circular tubular stent of other self-expandable valves. To limit the introduction of possible confounding factors in the analysis, the investigators decided on purpose not to include the Acurate in the present study.

Indication for TAVI respects international guidelines (EACTS 2017 Guidelines for Treatment of Valvular Heart Disease). A transthoracic examination is performed before the procedure at hospital admission. The in-hospital pathway pf examination is equal to every other patient treated in the participating centers.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 y.o.;
* The patient has undergone a previous TAVI;
* The Transcatheter Heart Valve (THV) implanted for TAVI procedure is a cumbersome and long self-expandable device (e.g. CoreValve, CoreValve Evolut R, Portico valve);
* The patient has already undergone a post-TAVI cardiac-gated CT-scan with contrast medium which includes the aortic arch (generally for other reasons such as participation into a clinical study with a previous Ethical Committee approval; residual aortic regurgitation assessment for Valve-in-Valve evaluation; TAVI complication assessment)

Exclusion Criteria:

* Age<18 y.o.;
* The Transcatheter Heart Valve (THV) implanted for TAVI procedure is a low-profile balloon-expandable device (e.g. Sapien);
* The patient has already undergone a post-TAVI cardiac-gated CT-scan with contrast medium which DOES NOT include the aortic arch.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: TAVI patients treated with a low-profile transcatheter aortic valve bioprosthesis
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2019-10-05 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
anatomical feasibility of surgical aortic cross-clamp and aortotomy after TAVI based on post-TAVI computed tomographies (CT). | up to 11 years
  evaluation at CT scan

CONTACTS AND LOCATIONS:
Locations (3):
- Rigshospitalet University Hospital - Cardiology Department, Copenhagen, Denmark
- Semmelweiss University - Cardiology Departmend, Budapest, Hungary
- IRCCS Ospedale San Raffaele - Cardiac Surgery Department, Milan, Italy

IPD SHARING:
Plan to Share IPD: No